CLINICAL TRIAL: NCT03902717
Title: An Observational Cohort Study to Investigate Patient-centered and Clinical Outcomes After Minimally Invasive Cardiothoracic Surgery
Brief Title: Patient-centered and Clinical Outcomes After Minimally Invasive Cardiothoracic Surgery
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Anesthesiologist, MD, PhD, Jessa Hospital
Other Study IDs: 18.47/ANESTH18.04
Record Dates: First submitted 2019-03-28; First posted 2019-04-04 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Disease; Surgery
Keywords: Minimally invasive cardiac surgery; Endoscopic coronary artery bypass grafting
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- minimally invasive cardiac surgery: Group of patients that will undergo minimally invasive cardiac surgery
  Interventions: Procedure: Minimally invasive cardiac surgery

INTERVENTIONS:
Procedure: Minimally invasive cardiac surgery — Patients will undergo minimally invasive cardiac surgery

SUMMARY:
Nowadays, minimally invasive cardiothoracic surgery techniques are being performed to treat patients with coronary heart diseases. These newly developed procedures include laparoscopic techniques that do not require median sternotomy, which has several beneficial effects for both patient and the hospital. Although retrospective data show promising results with respect to clinical outcomes (e.g. 30-day mortality rate, intensive care unit length of stay), no prospective data with respect to patient centered outcomes (e.g. quality of recovery, quality of life) are available yet. Therefore, the aim of this observational prospective study is to explore several patient centered and clinical outcomes of patients that are treated with these newly developed minimally invasive cardiac procedures. The comparative group consists of patients undergoing open CABG (invasive) and patients undergoing a Transcatheter Aortic Valve Implantation (TAVI).

DETAILED DESCRIPTION:
Introduction:

Coronary artery disease is a leading cause of adult mortality worldwide. One of the most commonly performed surgical interventions to treat this vascular disease is a myocardial revascularization, mostly performed via a Coronary Artery Bypass Graft (CABG) (1). Over time, new developments in cardiac surgery have led to the introduction of less invasive and minimally invasive cardiac procedures (2). These minimally invasive cardiac procedures are proven to be safe and feasible (3) and have excellent outcomes (4) (5) (6). More specifically, the short term outcomes include a reduced patient recovery time (5), lower transfusion rates, wound infections, hospitalization time and hospital mortality rate (4), while the long term outcomes comprise a better vessel graft patency (7) (8). Over the past few years, new minimally invasive cardiothoracic surgery techniques have been developed and are currently being implemented at the department of cardiothoracic surgery from the Jessa Hospital (e.g. endo-CABG, VATS Mitral, hybrid revascularization, Yil AVR). These newly developed procedures include laparoscopic techniques that do not require median sternotomy, which has several beneficial effects for both patient and the hospital. Also, these techniques allow a coronary revascularization or mitral valve repair or replacement without the use of expensive robotic equipment and exclusion of specific patients based on comorbidities (e.g. elderly patients, diabetic and/or obese patients). Currently, patients undergo cardiothoracic surgery via these techniques and although retrospective data from our hospital show promising results with respect to clinical outcomes (e.g. 30-day mortality rate, intensive care unit length of stay), no prospective data with respect to patient centered outcomes (e.g. quality of recovery, quality of life) are available yet. Therefore, the aim of this study is to explore several patient centered and clinical outcomes of patients that are treated with these newly developed minimally invasive cardiac procedures.The comparative group consists of patients undergoing open CABG (invasive) and patients undergoing a Transcatheter Aortic Valve Implantation (TAVI).

Outcome measures:

The goal of this study is to assess several patient central outcomes (e.g. quality of recovery measured with quality of life) and clinical outcomes (e.g. mortality rate, serious complications, major cardiac events, time registration in icu and hospital, duration of surgery, occlusion and perfusion time, surgical parameters, revalidation of the patients) after minimally invasive cardiothoracic surgery.

Design:

This study is a single-center prospective observational cohort study in which eligible patients that are treated via minimally invasive cardiac surgery will be included. Inclusion will last for 1 year and patients will be followed-up for 12 months.

Study Procedures:

After signing the informed consent form, the baseline tests will be performed the day before the surgery. On the day of the surgery, several surgical parameters will be measured as well as several parameters that are included in the standard clinical practice. 2 weeks, 1 month, 3 months and 1 year after the surgery, the QoL will be measured. Patient satisfaction will be assessed 3 months after surgery.

Statistical analysis:

Descriptive statistics will be presented as frequencies and percentages of the total amount of patients for categorical variables, while numerical variables will be presented as mean with variances. Results of the different questionnaires will be calculated according to their specific guidelines. The clinical significance of the questionnaires will be calculated via an effect size. A p-value <0.05 is considered statistical significant, while p<0.10 is considered a tendency.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Patients planned to undergo minimally invasive cardiac surgery by the following techniques:

  * Endo-CABG
  * Hybrid approach
  * VATS Mitral
  * Mini AVR
  * Yil AVR or open CABG or TAVI

Exclusion Criteria:

* Patients < 18 years old
* Patients that are not eligible to undergo minimally invasive cardiac surgery
* Patients that participate in other clinical, pharmaceutical or medical devices trials
* Patients that previously had a minimally invasive cardiac surgery and are now scheduled for a revision
* Patients that need a conversion to sternotomy or other non-minimally invasive technique
* Inability to understand and adhere to the study design

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are scheduled to undergo minimally invasive cardiac surgery, open CABG or TAVI
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | 1 month after surgery
  Quality of Recovery will be assessed via 2 questionnaires: the SF-36 and EQ-5D questionnaire concerning mobility, selfcare, daily activities and pain

SECONDARY OUTCOMES:
Quality of Recovery | 2 weeks after surgery
  Quality of Recovery will be assessed via 2 questionnaires: the SF-36 and EQ-5D questionnaire concerning mobility, selfcare, daily activities and pain
Quality of Recovery | 3 months after surgery
  Quality of Recovery will be assessed via 2 questionnaires: the SF-36 and EQ-5D questionnaire concerning mobility, selfcare, daily activities and pain
Quality of Recovery | 12 months after surgery
  Quality of Recovery will be assessed via 2 questionnaires: the SF-36 and EQ-5D questionnaire concerning mobility, selfcare, daily activities and pain
Routine measurements of standard medical practice | 12 months after surgery
  Routine measurements during and after surgery (e.g. amount of blood loss, time of ventilation, time of perfusion, hematology/blood chemistry, registration of mortality rates and complications after surgery, length of stay at the ICU department after surgery, length of stay in the hospital)
Patient satisfaction with respect to surgery | 3 months after surgery
  Patient satisfaction after surgery (assessed via the 7-point likert scale, with 1 being completely dissatisfied and 7 completely satisfied)
Physical recovery of patients after surgery | 2 weeks after surgery
  A maximal exercise test will be performed after surgery to asses revalidation of the patients
Physical recovery of patients after surgery | 1 month after surgery
  A maximal exercise test will be performed after surgery to asses revalidation of the patients
Physical recovery of patients after surgery | 3 months after surgery
  A maximal exercise test will be performed after surgery to asses revalidation of the patients
Physical recovery of patients after surgery | 12 months after surgery
  A maximal exercise test will be performed after surgery to asses revalidation of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Björn Stessel, MD, PhD, Principal Investigator — Jessa hospital, Hasselt
Locations (2):
- Belgium (2):
  - Jessa Hospital, Hasselt, Limburg
  - Department of Anesthesiology and Intensive Care, Hasselt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezelsoy M, Caynak B, Bayram M, Oral K, Bayramoglu Z, Sagbas E, Aytekin V, Akpinar B. The Comparison between Minimally Invasive Coronary Bypass Grafting Surgery and Conventional Bypass Grafting Surgery in Proximal LAD Lesion. Heart Surg Forum. 2015 Apr 28;18(2):E042-6. doi: 10.1532/hsf.1239. PMID 25924029
- [Background] Diodato M, Chedrawy EG. Coronary artery bypass graft surgery: the past, present, and future of myocardial revascularisation. Surg Res Pract. 2014;2014:726158. doi: 10.1155/2014/726158. Epub 2014 Jan 2. PMID 25374960
- [Background] Ruel M, Shariff MA, Lapierre H, Goyal N, Dennie C, Sadel SM, Sohmer B, McGinn JT Jr. Results of the Minimally Invasive Coronary Artery Bypass Grafting Angiographic Patency Study. J Thorac Cardiovasc Surg. 2014 Jan;147(1):203-8. doi: 10.1016/j.jtcvs.2013.09.016. Epub 2013 Oct 30. PMID 24183338
- [Background] Lapierre H, Chan V, Sohmer B, Mesana TG, Ruel M. Minimally invasive coronary artery bypass grafting via a small thoracotomy versus off-pump: a case-matched study. Eur J Cardiothorac Surg. 2011 Oct;40(4):804-10. doi: 10.1016/j.ejcts.2011.01.066. Epub 2011 Mar 9. PMID 21393011
- [Background] Poston RS, Tran R, Collins M, Reynolds M, Connerney I, Reicher B, Zimrin D, Griffith BP, Bartlett ST. Comparison of economic and patient outcomes with minimally invasive versus traditional off-pump coronary artery bypass grafting techniques. Ann Surg. 2008 Oct;248(4):638-46. doi: 10.1097/SLA.0b013e31818a15b5. PMID 18936577
- [Background] McGinn JT Jr, Usman S, Lapierre H, Pothula VR, Mesana TG, Ruel M. Minimally invasive coronary artery bypass grafting: dual-center experience in 450 consecutive patients. Circulation. 2009 Sep 15;120(11 Suppl):S78-84. doi: 10.1161/CIRCULATIONAHA.108.840041. PMID 19752390
- [Background] Biglioli P, Antona C, Alamanni F, Parolari A, Toscano T, Pompilio G, Polvani G. Minimally invasive direct coronary artery bypass grafting: midterm results and quality of life. Ann Thorac Surg. 2000 Aug;70(2):456-60. doi: 10.1016/s0003-4975(00)01371-0. PMID 10969662